CLINICAL TRIAL: NCT04206605
Title: A Phase 3, Multicenter, Randomized, Placebo-controlled, Double-blind Study to Evaluate the Efficacy and Safety of Lanadelumab for Prevention Against Acute Attacks of Non-histaminergic Angioedema With Normal C1-Inhibitor (C1-INH)
Brief Title: A Study of Lanadelumab in Teenagers and Adults to Prevent Acute Attacks of Non-histaminergic Angioedema With Normal C1-Inhibitor (C1-INH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHP643-303; 2019-001703-20 (EudraCT Number); jRCT2061210013 (Registry Identifier: Japan Ministry of Health, Labour and Welfare)
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Results first posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Angioedema
Keywords: Drug Therapy
MeSH Terms: conditions — Angioedema | interventions — lanadelumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo-matching lanadelumab subcutaneous (SC) injection once every 2 weeks (q2w) for up to 7 months.
  Interventions: Other: Placebo
- Lanadelumab 300mg (Experimental): Participants received 300 mg of lanadelumab solution in a prefilled syringe (PFS) as SC injection once (q2w) for up to 6 months.
  Interventions: Drug: Lanadelumab

INTERVENTIONS:
Other: Placebo — Placebo-matching lanadelumab SC injection.
  Arms: Placebo
Drug: Lanadelumab — Lanadelumab solution in a PFS for injection.
  Other Names: SHP643; DX-2930; TAK-743
  Arms: Lanadelumab 300mg

SUMMARY:
The main aim of this study is to check if repeated subcutaneous (SC) injections of lanadelumab can prevent angioedema attacks in teenagers and adults with non-histaminergic angioedema with normal C1-INH. Another aim is to check if they tolerate the repeated SC injections.

Participants will receive a SC injection of lanadelumab every two weeks for 26 weeks. The first two doses of lanadelumab will be given at the study clinic. Once a participant (and/or parent/caregiver) has been appropriately trained, lanadelumab can be self-injected. Visits to the study clinic are planned for the first, third and fourth week and then every 4 weeks.

DETAILED DESCRIPTION:
This study consists of non-histaminergic normal C1-INH angioedema population with 12 years of age and above. Participants will be randomized 2:1 to receive repeated SC administrations of lanadelumab or placebo in a double-blind fashion. Randomization will be stratified based on baseline angioedema attack rate (1 to less than (<) 2 attacks/4 weeks, and greater than (>=) 2 attacks/4 weeks), as well as subtype (known mutations, family history and unknown mutation, idiopathic).

ELIGIBILITY:
Inclusion Criteria:

The Participant will not be considered eligible for the study without meeting all of the applicable population criteria below.

* Males and females, 12 years of age and older for participants with non-histaminergic normal C1-INH angioedema at the time of signing of the informed consent form (ICF).
* Documented clinical history of recurrent attacks of angioedema in the absence of wheals/urticaria.
* Investigator-confirmed diagnosis of non-histaminergic bradykinin-mediated angioedema with normal C1-INH as documented by a history of angioedema attack(s) at screening and occurrence of attacks during the observation period:

  * History of recurrent angioedema with at least an average of 1 angioedema attack per 4 weeks prior to screening and this attack rate must be confirmed during the observation period while treated with chronic high-dose antihistamine (cetirizine 40 milligram per day [mg/day] or equivalent high-dose second-generation antihistamine medication).
  * Diagnostic testing results obtained during screening from a sponsor-approved central laboratory that confirm C1-INH function >= 50 percent (%) of normal and C4 level not below the normal range. With prior sponsor approval, participants may be retested during the observation period if results are incongruent with clinical history.
  * Clinical history of not responding to high-dose antihistamine treatment (cetirizine 40 mg/day or equivalent high-dose second-generation antihistamine medication), which must be confirmed during the observation period with at least 1 angioedema attack per 4 weeks with chronic high-dose antihistamine treatment and no significant difference (as assessed by the investigator and in consultation with the sponsor's medical monitor, as necessary) from the historic attack rate without high-dose antihistamine treatment.
* Agree to adhere to the protocol-defined schedule of treatments, assessments, and procedures.
* Participants >= 18 years of age must be willing to use icatibant as the rescue medication during the observation and treatment period. During the observation period, participants need to be treated with icatibant for at least 2 angioedema attacks or at least 1 moderate or severe attack. In the opinion of the investigator, participants with no response to icatibant for acute angioedema attacks in the past medical history/screening, or no improvement or worsened attack severity 2 hours after icatibant treatment during the observation period (based on totality of assessments), will not be included. Note: For participants 12 to < 18 years of age, standard of care therapy per local protocols should be provided.
* Males, or non-pregnant, non-lactating females who are of child-bearing potential and who agree to be abstinent or agree to comply with the applicable contraceptive requirements of this protocol for the duration of the study. Female participants of childbearing potential must have a negative serum pregnancy test at screening and must be willing to undergo pregnancy tests throughout the study. Females of non-childbearing potential are defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months.
* The participants (or the participant's parent/legal guardian, if applicable) has provided written informed consent approved by the institutional review board/research ethics board/ethics committee (IRB/REB/EC).
* If the participants is an adult, be informed of the nature of the study and provide written informed consent before any study-specific procedures are performed.

OR

- If the participants is a minor (i.e. < 18 years of age), have a parent/legal guardian who is informed of the nature of the study provide written informed consent (i.e. permission) for the minor to participate in the study before any study-specific procedures are performed. Assent will be obtained from minor participants.

Exclusion Criteria

The participant will be excluded from the study if any of the following exclusion criteria are met.

* Concomitant diagnosis of Type I or Type II HAE, or recurrent angioedema associated with urticaria.
* Dosing with any investigational drug or exposure to an investigational device within 4 weeks prior to screening.
* Exposure to angiotensin-converting enzyme (ACE) inhibitors or rituximab within 6 months prior to screening.
* Use of any estrogen-containing medications with systemic absorption (such as oral contraceptives or hormonal replacement therapy) within 4 weeks prior to screening.
* Response to omalizumab (prophylactic) or corticosteroid (acute/prophylactic) or epinephrine (acute) or anti-leukotrienes (prophylactic) treatments in the past.
* Use of long-term prophylactic therapy for HAE, e.g. C1-INH, attenuated androgens (e.g. danazol, methyltestosterone, testosterone), or anti-fibrinolytics within 2 weeks prior to entering the observation period as long as the investigator determines that doing so would not place the participant at any undue safety risk, and that the participant is at least 18 years of age.
* Any exposure to prophylactic plasma kallikrein inhibitors prior to screening.
* Use of short-term prophylaxis for HAE within 7 days prior to entering the observation period. Short-term prophylaxis is defined as C1-INH, attenuated androgens, or anti-fibrinolytics used to avoid angioedema complications from medically indicated procedures.
* Have any active infectious illness or fever defined as an oral temperature greater than (>) 38°C (100.4°F), tympanic > 38.5°C (101.3°F), axillary > 38°C (100.4°F), or rectal/core > 38.5°C (101.3°F) within 24 hours prior to the first dose of study drug in the treatment period.
* Any of the following liver function test abnormalities: alanine aminotransferase (ALT) > 3x upper limit of normal, or aspartate aminotransferase (AST) > 3x upper limit of normal, or total bilirubin > 2x upper limit of normal (unless the bilirubin elevation is a result of Gilbert's syndrome).
* Pregnancy or breast feeding.
* Participant has a known hypersensitivity to the investigational product or its components.
* Have any uncontrolled underlying medical condition which would require treatment adjustment during the study treatment period that, in the opinion of the investigator or sponsor, may confound the results of the safety assessments or may place the participant at risk. Participants with stable treatment for at least 3 months prior to screening and NOT expecting any change to their treatment regimen for 6 months during the study treatment period, will not be excluded.
* Have any condition (surgical or medical) that, in the opinion of the investigator or sponsor, may compromise their safety or compliance, preclude the successful conduct of the study, or interfere with interpretation of the results (e.g. significant pre-existing illness or other major comorbidities that the investigator considers may confound the interpretation of study results).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (45):
- United States (20):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Medical Research of Arizona, Scottsdale, Arizona
  - University of California San Diego, San Diego, California
  - AIRE Medical of Los Angeles, Santa Monica, California
  - Allergy and Asthma Clinical Research Inc, Walnut Creek, California
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - University of South Florida Asthma, Allergy & Immunology, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Kanarek Allergy, Asthma and Immunology, Overland Park, Kansas
  - Institute for Asthma & Allergy - Chevy Chase, Chevy Chase, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Jay M Kashkin, MD Allergy, Asthma and Immunology, Fair Lawn, New Jersey
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Optimed Research, LTD, Columbus, Ohio
  - Tanner Clinic, Layton, Utah
  - Seattle Allergy & Asthma Research Institute, Seattle, Washington
- Canada (2):
  - Ottawa Allergy Research Corporation, Ottawa, Ontario
  - Clinique Specialisee en Allergie de la Capitale, Québec, Quebec
- France (2):
  - CHU Grenoble Alpes, service de médecine interne, bureau de recherche clinique, Isere
  - Service médecine interne, hôpital Saint Antoine, Paris
- Germany (4):
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt am Main, Hesse
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz, Rhineland-Palatinate
  - Universitaetsklinikum Leipzig AoeR, Leipzig, Saxony
  - Klinikum rechts der Isar der TUM, HNO Klinik und Poliklinik, Munich
- Semmelweis Egyetem, Budapest, Hungary
- Italy (3):
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli (Presidio Ospedale Sacco), Milan
  - DAI di Medicina Interna, Immunologia Clinica, Patologia Clinica, Malattie Infettive, Napoli
  - Azienda Ospedaliera Universitaria OO. RR. S. Giovanni di Dio e Ruggi D'Aragona, Salerno
- Japan (2):
  - Hiroshima University Hospital, Hiroshima
  - Kobe University Hospital, Hyōgo
- Netherlands (3):
  - Amsterdam UMC, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - UMC Utrecht, Utrecht
- Poland (2):
  - NZOZ Homeo Medicus, Poradnia Alergologiczna, Bialystok
  - "ALL-MED" Specjalistyczna Opieka Medyczna Medyczny Instytut Badawczy, Wroclaw
- Spain (6):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Complexo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Riedl MA, Staubach P, Farkas H, Zanichelli A, Ren H, Nurse C, Andresen I, Juethner S, Yu M, Zhang J. Lanadelumab for prevention of attacks of non-histaminergic normal C1 inhibitor angioedema: results from the randomized, double-blind CASPIAN Study and CASPIAN open-label extension. Front Immunol. 2025 May 21;16:1502325. doi: 10.3389/fimmu.2025.1502325. eCollection 2025. PMID 40469312
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fdc4db2bf003ab47309

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 34 investigative sites in Canada, United States, Germany, Hungary, Italy, Spain, France, Japan, Netherlands, and Poland from 04 May 2020 to 20 October 2022.
Pre-assignment Details: Participants with a diagnosis of non-histaminergic angioedema were randomized in a 2:1 ratio to receive lanadelumab or placebo.
Groups:
- Placebo: Participants received placebo-matching lanadelumab subcutaneous (SC) injection once every 2 weeks (q2w) for up to 26 weeks.
- Lanadelumab 300 mg: Participants received 300 mg of lanadelumab solution in a prefilled syringe (PFS) as SC injection once q2w for up to 26 weeks.
Period: Overall Study
Arm/Group | Placebo | Lanadelumab 300 mg
Started | 27 | 50
Steady State Full Analysis Set (SS-FAS) (SS-FAS included all randomized participants who received any exposure to the investigational product during the presumed steady state period (Day 70 through Day 182).) | 27 | 49
Completed | 26 | 49
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) included all participants who received any exposure to the investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lanadelumab 300 mg | Total
Number analyzed (Participants) | 27 | 50 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (10.77) | 42.3 (14.06) | 42.8 (12.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 43 | 62
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 9
  Not Hispanic or Latino | 24 | 43 | 67
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 24 | 44 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 1 | 4 | 5
  France | 0 | 1 | 1
  Germany | 1 | 2 | 3
  Hungary | 1 | 1 | 2
  Italy | 3 | 6 | 9
  Japan | 2 | 2 | 4
  Netherlands | 2 | 2 | 4
  Poland | 4 | 2 | 6
  Spain | 1 | 2 | 3
  United States | 12 | 28 | 40
Height [Mean (Standard Deviation); unit: centimeter] | 168.32 (9.779) | 166.09 (8.232) | 166.87 (8.807)
Weight [Mean (Standard Deviation); unit: kilogram] | 82.09 (22.701) | 82.04 (25.217) | 82.06 (24.213)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per squared meter] — BMI is calculated as [weight(kg)/height(m^2)].
  kilogram per squared meter | 28.88 (7.413) | 29.75 (9.127) | 29.44 (8.525)

OUTCOME MEASURES:

1. Primary Outcome: Number of Investigator-Confirmed Angioedema Attacks During the Treatment Period of Day 0 Through Day 182
Description: An angioedema attack was defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). Attack rate was calculated for each participant as the number of attacks occurring during the specified period divided by the number of days the participant contributed to the specified period multiplied by 28 days. Number of investigator-confirmed angioedema attacks during the treatment period of Day 0 through Day 182 was assessed.
Time Frame: Day 0 through Day 182
Population: Full Analysis Set (FAS) included all randomized participants who received any exposure to the investigational product (IP) during the treatment period (Day 0 through Day 182).
Measure: Mean (Standard Deviation); unit: attacks/month
Groups:
- Placebo: Participants received placebo-matching lanadelumab subcutaneous (SC) injection once q2w for up to 26 weeks.
Arm/Group | Placebo | Lanadelumab 300 mg
Number analyzed (Participants) | 27 | 50
attacks/month | 1.63 (1.357) | 2.17 (2.062)
Statistical Analysis 1: Comparison: Placebo vs Lanadelumab 300 mg; Test type: Superiority; p = 0.899, Chi-squared — P-value was from Wald-based chi-square test; unadjusted for multiple testing; Rate Ratio = 1.02, 95% CI 2-sided [0.71 to 1.47]

2. Secondary Outcome: Number of Participants Achieving Attack-Free Status During the Treatment Period of Day 0 Through Day 182
Description: An angioedema attack was defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). A participant was considered as attack free during a time period if the participant has no investigator-confirmed angioedema attacks during that time period. For participants who discontinue the study prior to completion of the analysis period, participants were classified as attack-free or not based on the observed contribution to the analysis period. Number of participants achieving attack-free status during the treatment period of day 0 through day 182 was assessed.
Time Frame: Day 0 through Day 182
Population: FAS included all randomized participants who receive any exposure to the IP during the treatment period (Day 0 through Day 182).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lanadelumab 300 mg
Number analyzed (Participants) | 27 | 50
Participants | 1 | 2
Statistical Analysis 1: Comparison: Placebo vs Lanadelumab 300 mg; Test type: Superiority; p = 1.000, Cochran-Mantel-Haenszel — P-value was from the corresponding Mantel-Haenszel estimate for the common risk difference from Cochran-Mantel-Haenszel (CMH) test; unadjusted for multiple testing; Risk Difference (RD) = 0.003, 95% CI 2-sided [-0.153 to 0.114]

3. Secondary Outcome: Number of Investigator-Confirmed Moderate or Severe Angioedema Attacks During the Treatment Period of Day 0 Through Day 182
Description: Angioedema attack was defined as symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of tongue, palate, uvula, or larynx). Overall severity of the participant's angioedema attack was determined by site using the following definitions: 1. Mild: Transient or mild discomfort; 2. Moderate: Mild to moderate limitation in activity some assistance needed; 3. Severe: Marked limitation in activity, assistance required. Attack rate was calculated for each participant as the number of attacks occurring during the specified period divided by number of days the participant contributed to the specified period multiplied by 28 days.
Time Frame: Day 0 Through Day 182
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: attacks/month
Arm/Group | Placebo | Lanadelumab 300 mg
Number analyzed (Participants) | 27 | 50
attacks/month | 1.10 (0.984) | 1.45 (1.711)
Statistical Analysis 1: Comparison: Placebo vs Lanadelumab 300 mg; Test type: Superiority; p = 0.852, Chi-squared — P-value was from Wald-based chi-square test; unadjusted for multiple testing; Rate Ratio = 0.96, 95% CI 2-sided [0.62 to 1.48]

4. Secondary Outcome: Number of Investigator-Confirmed Angioedema Attacks During the Presumed Steady State Period of Day 70 Through Day 182
Description: An angioedema attack was defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). Number of investigator-confirmed angioedema attacks during the presumed steady state period of day 70 through day 182 were assessed. Attack rate was calculated for each participant as the number of attacks occurring during the specified period divided by the number of days the participant contributed to the specified period multiplied by 28 days.
Time Frame: Day 70 through Day 182
Population: Steady State (SS)-FAS included all randomized participants who received any exposure to the investigational product during the presumed steady state period (Day 70 through Day 182).
Measure: Mean (Standard Deviation); unit: attacks/month
Arm/Group | Placebo | Lanadelumab 300 mg
Number analyzed (Participants) | 27 | 49
attacks/month | 1.37 (1.231) | 2.05 (2.211)
Statistical Analysis 1: Comparison: Placebo vs Lanadelumab 300 mg; Test type: Superiority; p = 0.660, Chi-squared — P-value was from Wald-based chi-square test; unadjusted for multiple testing; Rate Ratio = 1.10, 95% CI 2-sided [0.72 to 1.70]

5. Secondary Outcome: Number of Participants Achieving Attack-Free Status During the Presumed Steady State Period of Day 70 Through Day 182
Description: An angioedema attack was defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). A participant was considered as attack free during a time period if the participant has no investigator-confirmed angioedema attacks during that time period. For participants who discontinue the study prior to completion of the analysis period, participants were classified as attack-free or not based on the observed contribution to the analysis period. Number of participants achieving attack-free status during the presumed steady state period of day 70 through day 182 was assessed.
Time Frame: Day 70 through Day 182
Population: SS-FAS included all randomized participants who received any exposure to the investigational product during the presumed steady state period (Day 70 through Day 182).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lanadelumab 300 mg
Number analyzed (Participants) | 27 | 49
Participants | 4 | 3
Statistical Analysis 1: Comparison: Placebo vs Lanadelumab 300 mg; Test type: Superiority; p = 0.250, Cochran-Mantel-Haenszel — P-value was from the corresponding Mantel-Haenszel estimate for the common risk difference from CMH test; unadjusted for multiple testing; Risk Difference (RD) = -0.087, 95% CI 2-sided [-0.280 to 0.063]

6. Secondary Outcome: Number of Participants With Maximum Attack Severity During Treatment Period of Day 0 Through Day 182
Description: An angioedema attack was defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). Number of participants with maximum attack severity during treatment period of day 0 through day 182 was assessed. Angioedema attack severity was calculated per participant based on the severity categories as follows: No attack, Mild, Moderate, and Severe.
Time Frame: Day 0 through Day 182
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lanadelumab 300 mg
Number analyzed (Participants) | 27 | 50
Participants
  No Attack | 1 | 2
  Mild | 2 | 4
  Moderate | 17 | 17
  Severe | 7 | 27

7. Secondary Outcome: Number of Investigator-Confirmed Moderate or Severe Angioedema Attacks During the Presumed Steady State Period of Day 70 Through Day 182
Description: An angioedema attack was defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). Attack rate was calculated for each participant as the number of attacks occurring during the specified period divided by the number of days the participant contributed to the specified period multiplied by 28 days. Number of investigator-confirmed moderate or severe angioedema attacks during the presumed steady state period of day 70 through day 182 were assessed.
Time Frame: Day 70 through Day 182
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: attacks/month
Arm/Group | Placebo | Lanadelumab 300 mg
Number analyzed (Participants) | 27 | 49
attacks/month | 0.97 (1.013) | 1.35 (1.764)
Statistical Analysis 1: Comparison: Placebo vs Lanadelumab 300 mg; Test type: Superiority; p = 0.896, Chi-squared — P-value was from Wald-based chi-square test; unadjusted for multiple testing; Rate Ratio = 0.97, 95% CI 2-sided [0.58 to 1.61]

8. Secondary Outcome: Number of Participants With Maximum Attack Severity During Presumed Steady State Period of Day 70 Through Day 182
Description: An angioedema attack was defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). Number of participants with maximum attack severity during the presumed steady state period of day 70 through day 182 was assessed. Angioedema attack severity was calculated per participant based on the severity categories as follows: No attack, Mild, Moderate, and Severe.
Time Frame: Day 70 through Day 182
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lanadelumab 300 mg
Number analyzed (Participants) | 27 | 49
Participants
  No Attack | 4 | 3
  Mild | 5 | 5
  Moderate | 12 | 23
  Severe | 6 | 18

9. Secondary Outcome: Time to First Angioedema Attack After Day 0 Through Day 182
Description: The time to the first angioedema attack (days) after Day 0 for the efficacy evaluation period of Day 0 through Day 182 was calculated from the date and time of the first dose of lanadelumab for the efficacy evaluation period (Day 0 through Day 182) to the date and time of the first in angioedema attack after the first dose for the efficacy evaluation period of Day 0 through Day 182. Participants with attacks occurring were the events. Participants who discontinue/complete the study prior to having an angioedema attack were censored. The data is reported for baseline angioedema attack rate groups i.e. 1 to < 2 Attacks/Month and >=2 Attacks/Month.
Time Frame: Day 0 Through Day 182
Population: FAS included all randomized participants who receive any exposure to the IP during the treatment period (Day 0 through Day 182). Number analyzed are the number of participants with attacks occurring as events.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Lanadelumab 300 mg
Number analyzed (Participants) | 27 | 50
days
  1 to <2 Attacks/Month: number analyzed (Participants) | 4 | 5
  1 to <2 Attacks/Month | 10.5 [6.6 to NA] — Upper limit of confidence Interval (CI) was not estimable due to insufficient number of participants with events. | 81.0 [6.4 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events.
  >=2 Attacks/Month: number analyzed (Participants) | 22 | 43
  >=2 Attacks/Month | 6.8 [1.4 to 11.6] | 5.9 [3.7 to 11.6]
Statistical Analysis 1: Comparison: Placebo vs Lanadelumab 300 mg; Test type: Superiority; p = 0.498, Log Rank — P-value comparing lanadelumab to placebo was from a log rank test stratified by baseline strata

10. Secondary Outcome: Time to First Angioedema Attack After Day 70 Through Day 182
Description: The time to the first angioedema attack (days) after Day 0 for the efficacy evaluation period of Day 70 through Day 182 was calculated from the date and time of the first dose of lanadelumab for the efficacy evaluation period (Day 70 through Day 182) to the date and time of the first in angioedema attack after the first dose for the efficacy evaluation period of Day 70 through Day 182. Participants with attacks occurring were the events. Participants who discontinue/complete the study prior to having an angioedema attack were censored. The data is reported for baseline angioedema attack rate groups i.e. 1 to < 2 Attacks/Month and >=2 Attacks/Month.
Time Frame: Day 70 through Day 182
Population: SS-FAS included all randomized participants who received any exposure to the investigational product during the presumed steady state period (Day 70 through Day 182). Number analyzed are the number of participants with attacks occurring as events.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Lanadelumab 300 mg
Number analyzed (Participants) | 27 | 49
days
  1 to <2 Attacks/Month: number analyzed (Participants) | 4 | 5
  1 to <2 Attacks/Month | 12.3 [10.3 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events. | 40.8 [3.4 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events.
  >=2 Attacks/Month: number analyzed (Participants) | 19 | 41
  >=2 Attacks/Month | 16.9 [6.7 to 32.5] | 10.6 [5.0 to 15.9]
Statistical Analysis 1: Comparison: Placebo vs Lanadelumab 300 mg; Test type: Superiority; p = 0.184, Log Rank — P-value comparing lanadelumab to placebo was from a log rank test stratified by baseline strata

11. Secondary Outcome: Number of Participants Achieving at Least 50 %, 70%, 90% and 100% Reduction in the Investigator-Confirmed Normalized Number of Attacks (NNA) Per 4 Weeks During Each of the Efficacy Evaluation Periods Relative to the Observation Period NNA
Description: The normalized number of investigator-confirmed angioedema attacks (NNA) during each efficacy evaluation period was expressed as a monthly (28 days) angioedema attack rate. Attack rate was calculated for each participant as the number of attacks occurring during the specified period divided by the number of days the participant contributed to the specified period multiplied by 28 days. Number of participants achieving at least 50 percent (%), 70%, 90% and 100% reduction in the investigator-confirmed normalized number of attacks per 4 weeks during each of the efficacy evaluation periods relative to the observation period NNA was assessed. The percentage reduction groups are not mutually exclusive, participants may appear in more than one group as applicable based on their percentage reduction.
Time Frame: Day 0 Through Day 182
Population: FAS included all randomized participants who receive any exposure to the IP during the treatment period (Day 0 through Day 182). Overall number of participants analyzed are the number of participants achieving at Least 50 %, 70%, 90% and 100% reduction in the investigator-confirmed normalized number of attacks.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lanadelumab 300 mg
Number analyzed (Participants) | 26 | 48
Participants
  >=50% Reduction | 13 | 28
  >=70% Reduction | 9 | 12
  >=90% Reduction | 3 | 6
  100% Reduction | 1 | 2

12. Secondary Outcome: Number of Participants Achieving Normalized Number of Attacks (NNA) Less Than (<)1.0 Per 4 Weeks During Each of the Efficacy Evaluation Periods
Description: The normalized number of investigator-confirmed angioedema attacks (NNA) during each efficacy evaluation period was expressed as a monthly (28 days) angioedema attack rate. Attack rate was calculated for each participant as the number of attacks occurring during the specified period divided by the number of days the participant contributed to the specified period multiplied by 28 days. Number of participants achieving normalized number of attacks < 1.0 per 4 weeks during each of the efficacy evaluation periods was assessed. The percentage reduction groups are not mutually exclusive, participants may appear in more than one group as applicable based on their percentage reduction.
Time Frame: Day 0 through Day 182, Day 70 through Day 182
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Groups:
- Lanadelumab 300 mg: Participants received 300 mg of lanadelumab solution in a prefilled syringe (PFS) as SC injection once q2w) for up to 26 weeks.
Arm/Group | Placebo | Lanadelumab 300 mg
Number analyzed (Participants) | 27 | 49
Participants
  >=50% Reduction | 14 | 31
  >=70% Reduction | 12 | 18
  >=90% Reduction | 5 | 5
  100% Reduction | 4 | 3

13. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Including Adverse Events of Special Interest (AESI) and Serious Adverse Events (SAEs)
Description: TEAE was defined as any event emerging or manifesting at or after the initiation of treatment with an investigational product (IP) or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the IP or medicinal product. SAE=untoward clinical manifestation of signs, symptoms or outcomes (whether considered related to investigational product or not and at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, congenital abnormality/birth defect, an important medical event. AESI included hypersensitivity reactions, events of disordered coagulation such as bleeding AESI, hypercoagulable AESI.
Time Frame: From the first study drug administration up to follow-up (Day 196)
Population: SAS included all participants who received any exposure to the IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lanadelumab 300 mg
Number analyzed (Participants) | 27 | 50
Participants
  Any TEAE | 23 | 46
  AESI | 0 | 1
  SAE | 1 | 7

14. Secondary Outcome: Plasma Concentrations of Lanadelumab
Time Frame: Pre-dose and post-dose at Days 0, 4, 14, 28, 56, 84, 112, 140, 168 and 182
Population: Pharmacokinetic Set (PK Set) included all participants in the SAS who had at least 1 evaluable postdose PK concentration value. Overall number of participants analyzed is the number of participants available with data for analyses. Number analyzed is the number of participants available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Placebo | Lanadelumab 300 mg
Number analyzed (Participants) | 27 | 49
nanogram/milliliter (ng/mL)
  Baseline: number analyzed (Participants) | 22 | 45
  Baseline | 661.573 (2991.1363) | 1.665 (7.8812)
  Day 0: number analyzed (Participants) | 0 | 1
  Day 0 |  | 0.000 (NA) — The standard deviation (SD) was not estimable for a single participant.
  Day 4: number analyzed (Participants) | 7 | 7
  Day 4 | 42.749 (113.1021) | 16895.996 (8136.5164)
  Day 14: number analyzed (Participants) | 16 | 32
  Day 14 | 5.366 (21.4650) | 11030.519 (4632.9383)
  Day 28: number analyzed (Participants) | 26 | 46
  Day 28 | 6.188 (17.9944) | 15969.813 (7210.5963)
  Day 56: number analyzed (Participants) | 27 | 46
  Day 56 | 16.820 (61.3021) | 20722.131 (8396.5980)
  Day 84: number analyzed (Participants) | 26 | 49
  Day 84 | 7.335 (30.0848) | 22698.616 (8953.3488)
  Day 112: number analyzed (Participants) | 25 | 48
  Day 112 | 5.604 (22.1843) | 22938.312 (10021.8340)
  Day 140: number analyzed (Participants) | 26 | 46
  Day 140 | 3.200 (16.3188) | 22778.286 (9680.4686)
  Day 168: number analyzed (Participants) | 24 | 48
  Day 168 | 9.260 (23.0763) | 21369.818 (11072.0806)
  Day 182: number analyzed (Participants) | 26 | 49
  Day 182 | 4.733 (18.7014) | 20496.158 (10774.2169)

15. Secondary Outcome: Plasma Kallikrein (pKal) Activity
Description: Plasma Kallikrein activity was measured by biomarker cleaved high molecular weight kininogen (cHMWK ) level to assess pharmacodynamics of lanadelumab.
Time Frame: Pre-dose and post-dose at Days 4, 14, 28, 56, 84, 112, 140, 168 and 182
Population: The Pharmacodynamic Set (PD Set) included all participants in the SAS who had at least 1 evaluable PD concentration value. Overall number of participants analyzed are the number of participants with data available for analyses. Number analyzed is the number of participants available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: % cHMWK
Arm/Group | Placebo | Lanadelumab 300 mg
Number analyzed (Participants) | 27 | 50
% cHMWK
  Baseline: number analyzed (Participants) | 25 | 50
  Baseline | 20.30 (14.927) | 18.69 (11.854)
  Day 4: number analyzed (Participants) | 7 | 7
  Day 4 | 25.94 (33.285) | 20.20 (20.333)
  Day 14: number analyzed (Participants) | 16 | 31
  Day 14 | 17.23 (9.801) | 12.83 (13.136)
  Day 28: number analyzed (Participants) | 27 | 47
  Day 28 | 16.16 (12.458) | 14.24 (13.472)
  Day 56: number analyzed (Participants) | 27 | 46
  Day 56 | 17.83 (12.169) | 15.88 (15.618)
  Day 84: number analyzed (Participants) | 27 | 48
  Day 84 | 17.00 (15.508) | 16.76 (15.941)
  Day 112: number analyzed (Participants) | 25 | 48
  Day 112 | 15.88 (11.109) | 16.12 (17.242)
  Day 140: number analyzed (Participants) | 27 | 47
  Day 140 | 17.40 (15.413) | 14.91 (14.656)
  Day 168: number analyzed (Participants) | 25 | 47
  Day 168 | 20.90 (16.588) | 15.07 (15.061)
  Day 182 | 18.08 (20.384) | 15.39 (15.333)

16. Secondary Outcome: Number of Participants With Neutralizing or Non-neutralizing Antidrug Antibodies (ADA) in Plasma
Description: Number of participants with neutralizing or non-neutralizing antidrug antibodies in plasma was assessed.
Time Frame: Pre-dose and post-dose at Days 28, 56, 84, 112, 140, 168 and 182
Population: FAS included all randomized participants who receive any exposure to the IP during the treatment period (Day 0 through Day 182). Number analyzed is the number of participants available for analyses at the given timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lanadelumab 300 mg
Number analyzed (Participants) | 27 | 50
Participants
  Baseline: number analyzed (Participants) | 22 | 46
  Baseline | 0 | 0
  Day 28: number analyzed (Participants) | 26 | 46
  Day 28 | 0 | 0
  Day 56: number analyzed (Participants) | 27 | 47
  Day 56 | 0 | 0
  Day 84: number analyzed (Participants) | 26 | 50
  Day 84 | 0 | 0
  Day 112: number analyzed (Participants) | 25 | 48
  Day 112 | 0 | 1
  Day 140: number analyzed (Participants) | 26 | 46
  Day 140 | 0 | 1
  Day 168: number analyzed (Participants) | 24 | 48
  Day 168 | 0 | 0
  Day 182: number analyzed (Participants) | 26 | 50
  Day 182 | 0 | 2

17. Secondary Outcome: Number of Participants With Change in Total Angioedema Quality of Life (AE-QoL) Questionnaire Score During the Treatment Period of Day 0 Through Day 182
Description: The AE-QoL questionnaire was a self-administered validated instrument to assess health related (HR) QoL among participants with recurrent angioedema. The AE-QoL consisted of 17 disease-specific quality-of-life items, to produce a total AEQoL score and 4 domain scores (functioning, fatigue/mood, fear/shame, and nutrition) and each of the 17 items has a five point response scale ranging from 0 (Never) to 4 (Very Often). The raw total score (mean of all item scores) was rescaled using linear transformations into final percentage scores ranging 0 to 100. Swelling episodes (SE); Trouble Concentrating (TC); Food and Beverages (F&B); negative effects (NE).
Time Frame: Baseline through Day 182
Population: SAS included all participants who receive any exposure to the IP. Overall number of participants analyzed are the number of participants with data available for analyses. Number analyzed is the number of participants available for analyses in the specific category.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lanadelumab 300 mg
Number analyzed (Participants) | 26 | 50
Participants
  Baseline: Work - Never: number analyzed (Participants) | 26 | 48
  Baseline: Work - Never | 7 | 6
  Baseline: Work - Rarely: number analyzed (Participants) | 26 | 48
  Baseline: Work - Rarely | 4 | 8
  Baseline: Work - Occasionally: number analyzed (Participants) | 26 | 48
  Baseline: Work - Occasionally | 6 | 14
  Baseline: Work - Often: number analyzed (Participants) | 26 | 48
  Baseline: Work - Often | 7 | 10
  Baseline: Work - Very Often: number analyzed (Participants) | 26 | 48
  Baseline: Work - Very Often | 2 | 10
  Baseline: Physical activity - Never: number analyzed (Participants) | 26 | 49
  Baseline: Physical activity - Never | 1 | 4
  Baseline: Physical activity - Rarely: number analyzed (Participants) | 26 | 49
  Baseline: Physical activity - Rarely | 1 | 7
  Baseline: Physical activity - Occasionally: number analyzed (Participants) | 26 | 49
  Baseline: Physical activity - Occasionally | 16 | 15
  Baseline: Physical activity - Often: number analyzed (Participants) | 26 | 49
  Baseline: Physical activity - Often | 4 | 12
  Baseline: Physical activity - Very Often: number analyzed (Participants) | 26 | 49
  Baseline: Physical activity - Very Often | 4 | 11
  Baseline: Leisure time - Never: number analyzed (Participants) | 26 | 49
  Baseline: Leisure time - Never | 1 | 4
  Baseline: Leisure time - Rarely: number analyzed (Participants) | 26 | 49
  Baseline: Leisure time - Rarely | 5 | 9
  Baseline: Leisure time - Occasionally: number analyzed (Participants) | 26 | 49
  Baseline: Leisure time - Occasionally | 12 | 17
  Baseline: Leisure time - Often: number analyzed (Participants) | 26 | 49
  Baseline: Leisure time - Often | 5 | 15
  Baseline: Leisure time - Very Often: number analyzed (Participants) | 26 | 49
  Baseline: Leisure time - Very Often | 3 | 4
  Baseline: Social relations - Never: number analyzed (Participants) | 26 | 49
  Baseline: Social relations - Never | 2 | 4
  Baseline: Social relations - Rarely: number analyzed (Participants) | 26 | 49
  Baseline: Social relations - Rarely | 4 | 9
  Baseline: Social relations - Occasionally: number analyzed (Participants) | 26 | 49
  Baseline: Social relations - Occasionally | 12 | 16
  Baseline: Social relations - Often: number analyzed (Participants) | 26 | 49
  Baseline: Social relations - Often | 7 | 16
  Baseline: Social relations - Very Often: number analyzed (Participants) | 26 | 49
  Baseline: Social relations - Very Often | 1 | 4
  Baseline: Eating and drinking - Never: number analyzed (Participants) | 26 | 49
  Baseline: Eating and drinking - Never | 3 | 8
  Baseline: Eating and drinking - Rarely: number analyzed (Participants) | 26 | 49
  Baseline: Eating and drinking - Rarely | 6 | 10
  Baseline: Eating and drinking - Occasionally: number analyzed (Participants) | 26 | 49
  Baseline: Eating and drinking - Occasionally | 9 | 16
  Baseline: Eating and drinking - Often: number analyzed (Participants) | 26 | 49
  Baseline: Eating and drinking - Often | 6 | 13
  Baseline: Eating and drinking - Very often: number analyzed (Participants) | 26 | 49
  Baseline: Eating and drinking - Very often | 2 | 2
  Baseline: Difficulty falling asleep - Never: number analyzed (Participants) | 26 | 49
  Baseline: Difficulty falling asleep - Never | 3 | 7
  Baseline: Difficulty falling asleep - Rarely: number analyzed (Participants) | 26 | 49
  Baseline: Difficulty falling asleep - Rarely | 3 | 7
  Baseline: Difficulty falling asleep - Occasionally: number analyzed (Participants) | 26 | 49
  Baseline: Difficulty falling asleep - Occasionally | 11 | 17
  Baseline: Difficulty falling asleep - Often: number analyzed (Participants) | 26 | 49
  Baseline: Difficulty falling asleep - Often | 5 | 8
  Baseline: Difficulty falling asleep - Very often: number analyzed (Participants) | 26 | 49
  Baseline: Difficulty falling asleep - Very often | 4 | 10
  Baseline: Wake up during the night - Never: number analyzed (Participants) | 26 | 49
  Baseline: Wake up during the night - Never | 2 | 2
  Baseline: Wake up during the night - Rarely: number analyzed (Participants) | 26 | 49
  Baseline: Wake up during the night - Rarely | 7 | 11
  Baseline: Wake up during the night - Occasionally: number analyzed (Participants) | 26 | 49
  Baseline: Wake up during the night - Occasionally | 5 | 12
  Baseline: Wake up during the night - Often: number analyzed (Participants) | 26 | 49
  Baseline: Wake up during the night - Often | 6 | 10
  Baseline: Wake up during the night - Very often: number analyzed (Participants) | 26 | 49
  Baseline: Wake up during the night - Very often | 6 | 14
  Baseline: Tired during the day - Never: number analyzed (Participants) | 26 | 49
  Baseline: Tired during the day - Never | 1 | 3
  Baseline: Tired during the day - Rarely: number analyzed (Participants) | 26 | 49
  Baseline: Tired during the day - Rarely | 7 | 8
  Baseline: Tired during the day - Occasionally: number analyzed (Participants) | 26 | 49
  Baseline: Tired during the day - Occasionally | 6 | 16
  Baseline: Tired during the day - Often: number analyzed (Participants) | 26 | 49
  Baseline: Tired during the day - Often | 7 | 9
  Baseline: Tired during the day - Very often: number analyzed (Participants) | 26 | 49
  Baseline: Tired during the day - Very often | 5 | 13
  Baseline: Trouble concentrating - Never: number analyzed (Participants) | 26 | 49
  Baseline: Trouble concentrating - Never | 2 | 3
  Baseline: Trouble concentrating - Rarely: number analyzed (Participants) | 26 | 49
  Baseline: Trouble concentrating - Rarely | 8 | 14
  Baseline: Trouble concentrating - Occasionally: number analyzed (Participants) | 26 | 49
  Baseline: Trouble concentrating - Occasionally | 10 | 14
  Baseline: Trouble concentrating - Often: number analyzed (Participants) | 26 | 49
  Baseline: Trouble concentrating - Often | 4 | 10
  Baseline: Trouble concentrating - Very often: number analyzed (Participants) | 26 | 49
  Baseline: Trouble concentrating - Very often | 2 | 8
  Baseline: Feel depressed - Never: number analyzed (Participants) | 26 | 49
  Baseline: Feel depressed - Never | 9 | 10
  Baseline: Feel depressed - Rarely: number analyzed (Participants) | 26 | 49
  Baseline: Feel depressed - Rarely | 5 | 18
  Baseline: Feel depressed - Occasionally: number analyzed (Participants) | 26 | 49
  Baseline: Feel depressed - Occasionally | 5 | 11
  Baseline: Feel depressed - Often: number analyzed (Participants) | 26 | 49
  Baseline: Feel depressed - Often | 6 | 7
  Baseline: Feel depressed - Very often: number analyzed (Participants) | 26 | 49
  Baseline: Feel depressed - Very often | 1 | 3
  Baseline: Limit your choices of food or beverages - Never: number analyzed (Participants) | 26 | 49
  Baseline: Limit your choices of food or beverages - Never | 10 | 17
  Baseline: Limit your choices of food or beverages - Rarely: number analyzed (Participants) | 26 | 49
  Baseline: Limit your choices of food or beverages - Rarely | 1 | 4
  Baseline: Limit your choices of food or beverages - Occasionally: number analyzed (Participants) | 26 | 49
  Baseline: Limit your choices of food or beverages - Occasionally | 2 | 13
  Baseline: Limit your choices of food or beverages - Often: number analyzed (Participants) | 26 | 49
  Baseline: Limit your choices of food or beverages - Often | 8 | 7
  Baseline: Limit your choices of food or beverages - Very often: number analyzed (Participants) | 26 | 49
  Baseline: Limit your choices of food or beverages - Very often | 5 | 8
  Baseline: Swelling episodes place a burden on you - Never: number analyzed (Participants) | 26 | 49
  Baseline: Swelling episodes place a burden on you - Never | 1 | 1
  Baseline: Swelling episodes place a burden on you - Rarely: number analyzed (Participants) | 26 | 49
  Baseline: Swelling episodes place a burden on you - Rarely | 1 | 0
  Baseline: Swelling episodes place a burden on you - Occasionally: number analyzed (Participants) | 26 | 49
  Baseline: Swelling episodes place a burden on you - Occasionally | 7 | 8
  Baseline: Swelling episodes place a burden on you - Often: number analyzed (Participants) | 26 | 49
  Baseline: Swelling episodes place a burden on you - Often | 10 | 24
  Baseline: Swelling episodes place a burden on you - Very often: number analyzed (Participants) | 26 | 49
  Baseline: Swelling episodes place a burden on you - Very often | 7 | 16
  Baseline: Swelling episode could occur suddenly - Never: number analyzed (Participants) | 26 | 49
  Baseline: Swelling episode could occur suddenly - Never | 1 | 2
  Baseline: Swelling episode could occur suddenly - Rarely: number analyzed (Participants) | 26 | 49
  Baseline: Swelling episode could occur suddenly - Rarely | 4 | 1
  Baseline: Swelling episode could occur suddenly - Occasionally: number analyzed (Participants) | 26 | 49
  Baseline: Swelling episode could occur suddenly - Occasionally | 4 | 12
  Baseline: Swelling episode could occur suddenly - Often: number analyzed (Participants) | 26 | 49
  Baseline: Swelling episode could occur suddenly - Often | 6 | 16
  Baseline: Swelling episode could occur suddenly - Very often: number analyzed (Participants) | 26 | 49
  Baseline: Swelling episode could occur suddenly - Very often | 11 | 18
  Baseline: Freq of swelling episodes might increase - Never: number analyzed (Participants) | 26 | 49
  Baseline: Freq of swelling episodes might increase - Never | 2 | 1
  Baseline: Freq of swelling episodes might increase - Rarely: number analyzed (Participants) | 26 | 49
  Baseline: Freq of swelling episodes might increase - Rarely | 3 | 3
  Baseline: Freq of swelling episodes might increase - Occasionally: number analyzed (Participants) | 26 | 49
  Baseline: Freq of swelling episodes might increase - Occasionally | 5 | 7
  Baseline: Freq of swelling episodes might increase - Often: number analyzed (Participants) | 26 | 49
  Baseline: Freq of swelling episodes might increase - Often | 8 | 21
  Baseline: Freq of swelling episodes might increase - Very often: number analyzed (Participants) | 26 | 49
  Baseline: Freq of swelling episodes might increase - Very often | 8 | 17
  Baseline: Ashamed to go out due to swell episodes - Never: number analyzed (Participants) | 26 | 49
  Baseline: Ashamed to go out due to swell episodes - Never | 6 | 10
  Baseline: Ashamed to go out due to swell episodes - Rarely: number analyzed (Participants) | 26 | 49
  Baseline: Ashamed to go out due to swell episodes - Rarely | 1 | 7
  Baseline: Ashamed to go out due to swell episodes - Occasionally: number analyzed (Participants) | 26 | 49
  Baseline: Ashamed to go out due to swell episodes - Occasionally | 8 | 10
  Baseline: Ashamed to go out due to swell episodes - Often: number analyzed (Participants) | 26 | 49
  Baseline: Ashamed to go out due to swell episodes - Often | 4 | 11
  Baseline: Ashamed to go out due to swell episodes - Very often: number analyzed (Participants) | 26 | 49
  Baseline: Ashamed to go out due to swell episodes - Very often | 7 | 11
  Baseline: Swelling episodes make you embarrassed - Never: number analyzed (Participants) | 26 | 49
  Baseline: Swelling episodes make you embarrassed - Never | 5 | 9
  Baseline: Swelling episodes make you embarrassed - Rarely: number analyzed (Participants) | 26 | 49
  Baseline: Swelling episodes make you embarrassed - Rarely | 4 | 5
  Baseline: Swelling episodes make you embarrassed - Occasionally: number analyzed (Participants) | 26 | 49
  Baseline: Swelling episodes make you embarrassed - Occasionally | 6 | 13
  Baseline: Swelling episodes make you embarrassed - Often: number analyzed (Participants) | 26 | 49
  Baseline: Swelling episodes make you embarrassed - Often | 3 | 8
  Baseline: Swelling episodes make you embarrassed - Very often: number analyzed (Participants) | 26 | 49
  Baseline: Swelling episodes make you embarrassed - Very often | 8 | 14
  Baseline: Afraid of long term negative effects - Never: number analyzed (Participants) | 26 | 49
  Baseline: Afraid of long term negative effects - Never | 3 | 9
  Baseline: Afraid of long term negative effects - Rarely: number analyzed (Participants) | 26 | 49
  Baseline: Afraid of long term negative effects - Rarely | 6 | 15
  Baseline: Afraid of long term negative effects - Occasionally: number analyzed (Participants) | 26 | 49
  Baseline: Afraid of long term negative effects - Occasionally | 6 | 4
  Baseline: Afraid of long term negative effects - Often: number analyzed (Participants) | 26 | 49
  Baseline: Afraid of long term negative effects - Often | 6 | 12
  Baseline: Afraid of long term negative effects - Very often: number analyzed (Participants) | 26 | 49
  Baseline: Afraid of long term negative effects - Very often | 5 | 9
  Day 182: Work - Never | 3 | 17
  Day 182: Work - Rarely | 10 | 8
  Day 182: Work - Occasionally | 8 | 12
  Day 182: Work - Often | 4 | 10
  Day 182: Work - Very Often | 1 | 3
  Day 182: Physical activity - Never | 3 | 13
  Day 182: Physical activity - Rarely | 10 | 12
  Day 182: Physical activity - Occasionally | 8 | 13
  Day 182: Physical activity - Often | 4 | 8
  Day 182: Physical activity - Very often | 1 | 4
  Day 182: Leisure time - Never | 3 | 14
  Day 182: Leisure time - Rarely | 12 | 15
  Day 182: Leisure time - Occasionally | 7 | 10
  Day 182: Leisure time - Often | 3 | 7
  Day 182: Leisure time - Very often | 1 | 4
  Day 182: Social relations - Never | 4 | 15
  Day 182: Social relations - Rarely | 8 | 11
  Day 182: Social relations - Occasionally | 9 | 13
  Day 182: Social relations - Often | 2 | 6
  Day 182: Social relations - Very often | 3 | 5
  Day 182: Eating and drinking - Never | 5 | 18
  Day 182: Eating and drinking - Rarely | 8 | 8
  Day 182: Eating and drinking - Occasionally | 8 | 9
  Day 182: Eating and drinking - Often | 4 | 14
  Day 182: Eating and drinking - Very often | 1 | 1
  Day 182: Difficulty falling asleep - Never | 4 | 9
  Day 182: Difficulty falling asleep - Rarely | 7 | 15
  Day 182: Difficulty falling asleep - Occasionally | 8 | 12
  Day 182: Difficulty falling asleep - Often | 6 | 9
  Day 182: Difficulty falling asleep - Very often | 1 | 5
  Day 182: Wake up during the night - Never | 1 | 9
  Day 182: Wake up during the night - Rarely | 7 | 10
  Day 182: Wake up during the night - Occasionally | 8 | 15
  Day 182: Wake up during the night - Often | 7 | 9
  Day 182: Wake up during the night - Very often | 3 | 7
  Day 182: Tired during the day - Never | 2 | 9
  Day 182: Tired during the day - Rarely | 6 | 15
  Day 182: Tired during the day - Occasionally | 11 | 12
  Day 182: Tired during the day - Often | 6 | 9
  Day 182: Tired during the day - Very often | 1 | 5
  Day 182: Trouble concentrating - Never | 2 | 13
  Day 182: Trouble concentrating - Rarely | 17 | 10
  Day 182: Trouble concentrating - Occasionally | 5 | 14
  Day 182: Trouble concentrating - Often | 1 | 10
  Day 182: Trouble concentrating - Very often | 1 | 3
  Day 182: Feel depressed - Never | 8 | 18
  Day 182: Feel depressed - Rarely | 8 | 18
  Day 182: Feel depressed - Occasionally | 5 | 7
  Day 182: Feel depressed - Often | 4 | 5
  Day 182: Feel depressed - Very often | 1 | 2
  Day 182: Limit your choices of food or beverages - Never | 7 | 19
  Day 182: Limit your choices of food or beverages - Rarely | 6 | 8
  Day 182: Limit your choices of food or beverages - Occasionally | 6 | 10
  Day 182: Limit your choices of food or beverages - Often | 5 | 8
  Visit 26: Limit your choices of food or beverages - Very often | 2 | 5
  Day 182: Swelling episodes place a burden on you - Never | 2 | 6
  Day 182: Swelling episodes place a burden on you - Rarely | 7 | 9
  Day 182: Swelling episodes place a burden on you - Occasionally | 8 | 17
  Day 182: Swelling episodes place a burden on you - Often | 7 | 7
  Day 182: Swelling episodes place a burden on you - Very often | 2 | 11
  Day 182: Swelling episode could occur suddenly - Never | 2 | 7
  Day 182: Swelling episode could occur suddenly - Rarely | 6 | 14
  Day 182: Swelling episode could occur suddenly - Occasionally | 9 | 10
  Day 182: Swelling episode could occur suddenly - Often | 5 | 7
  Day 182: Swelling episode could occur suddenly - Very often | 4 | 12
  Day 182: Freq of swelling episodes might increase - Never | 2 | 7
  Day 182: Freq of swelling episodes might increase - Rarely | 7 | 12
  Day 182: Freq of swelling episodes might increase - Occasionally | 9 | 13
  Day 182: Freq of swelling episodes might increase - Often | 5 | 6
  Day 182: Freq of swelling episodes might increase - Very often | 3 | 12
  Day 182: Ashamed to go out due to swell episodes - Never | 5 | 15
  Day 182: Ashamed to go out due to swell episodes - Rarely | 8 | 11
  Day 182: Ashamed to go out due to swell episodes - Occasionally | 4 | 10
  Day 182: Ashamed to go out due to swell episodes - Often | 7 | 8
  Day 182: Ashamed to go out due to swell episodes - Very often | 2 | 6
  Day 182: Swelling episodes make you embarrassed - Never | 7 | 14
  Day 182: Swelling episodes make you embarrassed - Rarely | 5 | 10
  Day 182: Swelling episodes make you embarrassed - Occasionally | 6 | 10
  Day 182: Swelling episodes make you embarrassed - Often | 6 | 8
  Day 182: Swelling episodes make you embarrassed - Very often | 2 | 8
  Day 182: Afraid of long term negative effects - Never | 4 | 15
  Day 182: Afraid of long term negative effects - Rarely | 10 | 13
  Day 182: Afraid of long term negative effects - Occasionally | 7 | 11
  Day 182: Afraid of long term negative effects - Often | 1 | 3
  Day 182: Afraid of long term negative effects - Very often | 4 | 8

ADVERSE EVENTS:
Time Frame: From start of the study up to follow up (Day 196)
Arm/Group | Placebo | Lanadelumab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/27 | 7/50
Other Adverse Events (participants affected / at risk) | 27/27 | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | Lanadelumab 300 mg (N=50)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (8)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | Lanadelumab 300 mg (N=50)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (8) | 4 (4)
Fatigue (General disorders) | 2 (9) | 4 (13)
Injection site erythema (General disorders) | 3 (6) | 3 (22)
Injection site pain (General disorders) | 7 (9) | 15 (61)
Pyrexia (General disorders) | 2 (2) | 3 (3)
COVID-19 (Infections and infestations) | 4 (4) | 3 (3)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (5)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (6)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (4)
Headache (Nervous system disorders) | 6 (13) | 6 (13)
Migraine (Nervous system disorders) | 1 (1) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Angioedema (Skin and subcutaneous tissue disorders) | 26 (305) | 48 (740)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/05/NCT04206605/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT04206605/SAP_001.pdf